CLINICAL TRIAL: NCT04620564
Title: Longitudinal Analysis of Mental Disorders, Psychosocial Distress and Psycho-oncological Care Needs of Patients and Their Relatives Stratified by Biopsychosocial Factors (LUPE)
Brief Title: Longitudinal Analysis of Mental Disorders, Psychosocial Distress and Care Needs of Patients and Their Relatives
Acronym: LUPE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Leipzig (Other)
Collaborators: Charite University, Berlin, Germany (Other); Hannover Medical School (Other); German Cancer Aid (Other)
Responsible Party: Principal Investigator, Anja Mehnert, Prof, University of Leipzig
Other Study IDs: DKH-70113544
Record Dates: First submitted 2020-10-05; First posted 2020-11-09 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Neoplasm Malignant
Keywords: psycho-oncology; psychological care; utilization; distress; mental disorders; neoplasm malignant; cancer
MeSH Terms: conditions — Neoplasms; Patient Acceptance of Health Care; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients
- Relatives

SUMMARY:
The primary objectives of this prospective observational multicenter study LUPE are to assess the prevalence of mental disorders according to the DSM-5 (objective need for psycho-oncological support), psychosocial distress, psycho-oncological care needs and utilization of psycho-oncological support services (subjective need for support) of cancer patients and their relatives during the first months of cancer survivorship stratified by biopsychosocial factors including socioeconomic status. The investigators further aim to identify moderating and mediating as well as associated factors for psychological distress and supportive care needs.

LUPE will include 2000 adult patients with solid tumor entities and one relative per patient at 4 measurement points from time of diagnosis to follow-up (+18 months) (t1: after diagnosis, t2: 6 month later, t3: 6 month later, t4: 6 month later).

The investigators aim to generate a quota sample according to socioeconomic status (SES) that is representative of the German overall population.

All participants will receive validated self-report questionnaires. Cancer patients will be interviewed using the standardized clinical interview SCID-5.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of malignant solid tumor
* a maximum time period after diagnosis of 4-8 weeks
* minimum age of 18 years
* cognitive ability to consent to study participation

Exclusion Criteria:

* presence of hematological cancers
* patients with cancer recurrence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid oncological tumors diagnosed no more than 4-8 weeks ago and meeting the inclusion criteria. The relatives of the patients do not have to meet any special inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of mental disorders according to the DSM-5 (objective need for psycho-oncological support) in cancer patients and the changes over time | after the diagnosis (up to 8 weeks) and at every follow up (Month 6, Month 12, Month 18)
  SCID (Structured Clinical Interview)
Frequency and extent of psychological distress (Depression) (subjective psycho-oncological support needs) in cancer patients and their relatives and the changes over time | after the diagnosis (up to 8 weeks) and at every follow up (Month 6, Month 12, Month 18)
  PHQ (Patient Health Questionnaire - Depression)
Frequency and extent of psychological distress (Anxiety) (subjective psycho-oncological support needs) in cancer patients and their relatives and the changes over time | after the diagnosis (up to 8 weeks) and at every follow up (Month 6, Month 12, Month 18)
  GAD (Generalized Anxiety Disorder)
Use of psycho-oncological support services by patients and relatives and the changes over time | after the diagnosis (up to 8 weeks) and at every follow up (Month 6, Month 12, Month 18)
Changes in Quality of Life and the changes over time | after the diagnosis (up to 8 weeks) and at every follow up (Month 6, Month 12, Month 18)
  EORTC (European Organisation for Research and Treatment of Cancer - Quality of life)

SECONDARY OUTCOMES:
Protective factors and stress-increasing risk factors within the dyad of relatives and the changes over time | after the diagnosis (up to 8 weeks) and at every follow up (Month 6, Month 12, Month 18)
  DCI (Dyadic Coping Inventar)

OTHER OUTCOMES:
Adherence of the patients | at follow up (Month 6)
  AAQ (Adherence Assessment Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Mehnert-Theuerkauf, Prof, Principal Investigator — Universitätsklinikum Leipzig
Locations (1):
- Department of Medical Psychology and Medical Sociology, University Medical Center Leipzig, Leipzig, Saxony, Germany

REFERENCES:
- [Derived] Mehnert-Theuerkauf A, Goerling U, Zimmermann T, Ernst J, Hermann M, Hornemann B, Keilholz U, Lordick F, Knesebeck OVD, Kissane D, Koditz AK, Springer F. Early Cancer Survivorship Distress Trajectories Associated With Socioeconomic Status and Age: Findings From a Multicenter Prospective Study. Cancer Med. 2025 Aug;14(15):e71076. doi: 10.1002/cam4.71076. PMID 40747744
- [Derived] Mehnert-Theuerkauf A, Hufeld JM, Esser P, Goerling U, Hermann M, Zimmermann T, Reuter H, Ernst J. Prevalence of mental disorders, psychosocial distress, and perceived need for psychosocial support in cancer patients and their relatives stratified by biopsychosocial factors: rationale, study design, and methods of a prospective multi-center observational cohort study (LUPE study). Front Psychol. 2023 Apr 20;14:1125545. doi: 10.3389/fpsyg.2023.1125545. eCollection 2023. PMID 37151329